CLINICAL TRIAL: NCT04517539
Title: Abscopal Effect of SBRT in Combination With rhGM-CSF and INF-α 2b for Metastatic Thymic Epithelial Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Cancer Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC-SGCI002
Record Dates: First submitted 2020-08-16; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Thymic Epithelial Tumor
MeSH Terms: conditions — Thymic epithelial tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT+GM-CSF+INF-αb (Experimental): Metastasis lesion will be treated with a SBRT of 30Gy/5F from day 1 to day 5 . Injection of Immunological Agenthuman recombined granulocyte-macrophage colony stimulating factor (125ug/m² per day) will be executed from day 1 to day 14 in this cycle.Subcutaneous injection of Peginterferon alfa-b2(90ug) will be executed in day8. Another metastasis lesion will be treated likewise concurrently with rhGM-CSF in a consecutive cycle. Injection of Peginterferon alfa-b2(90ug) will be executed in day8 of this cycle.
  Interventions: Drug: rhGM-CSF，Peginterferon alfa-b2，radiation

INTERVENTIONS:
Drug: rhGM-CSF，Peginterferon alfa-b2，radiation — Radiation:
  If there are two measurable lesions totally, One lesion received radiotherapy for 30 Gy in 5 fractions and rested for one week; If there are three measurable lesions totally, two lesion received radiotherapy for 30 Gy in 5 fractions separately.
  drug: Patients were injected subcutaneously rhGM-CSF 125mg/m2 per day from day1 to day 14, every three weeks, concurrent with radiotherapy. Peginterferon alfa-b2 90 ug in d8 in each cycle.
  And the 1 month after the end of all radiotherapy courses, 4 weeks as a course of treatment, once per course of treatment, each dose is 90μg until desease progress.

SUMMARY:
The purpose of this study is to determine whether stereotactic body radiotherapy (SBRT) combined with recombined human granulocyte-macrophage colony stimulating factor(rhGM-CSF) and Peginterferon alfa-2b is safe, effective in the treatment of patients with metastatic thymic epithelial tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Histologically proven Thymic epithelial tumors；
3. Stage IV according to UICC stage system(version 8,2017), at least with two evaluable abscopal lesions (≥1cm)（excluding intestinal metastasis）;
4. Evaluated as effective or stable disease after first-line chemotherapy or progressed after second-line chemotherapy (progression sites were no more than three sites);
5. ECOG performance status: 0-1;
6. Life expectancy ≥ 3 months.
7. Adequate baseline organ and marrow function: absolute neutrophil count greater than 1500 cells per μL, platelet concentration of greater than 50 000 per μL, total bilirubin less than 1•5 times the upper limit of normal (ULN), aspartate aminotransferase and alanine aminotransferase less than 2•5 times the ULN, and serum creatinine less than 1•5 times the ULN;
8. Female subjects have a negative urine or serum pregnancy test within 1 week prior to treatment if of childbearing potential;
9. Asymptomatic subjects with brain metastasis can be included, but the sites of brain cannot be considered as target sites;
10. Asymptomatic subjects with bone metastasis can be included, but the sites of bone cannot be considered as target sites.

Exclusion Criteria:

1. Having received immunotherapy within 4 weeks prior to inclusion;
2. Allergic to GM-CSF, INF-α2b or diagnosed with immune system disease, receiving immunosuppressant, such as prednisone, dexamethasone, methylprednisolone, methotrexate, hydroxychloroquine, cyclophosphamide, azathioprine and so one;
3. receiving treatment of other trials;
4. Any unstable systemic disease, including active infection, symptomatic congestive heart failure,myocardial infarction onset six months before included into the group, unstable angina, and severe arrhythmia, uncontrolled chronic lung disease;
5. unwilling to sign consent;
6. Women in pregnancy or lactation;
7. Other malignancy except for non-melanoma carcinoma of the skin or in situ carcinoma of the cervix.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
The abscopal effect rate | up to 12 months
  The proportion of patients with an abscopal response assessed after the initiation of treatment

SECONDARY OUTCOMES:
Progression free survival | up to 60 months
  From the date of enrollment to the date of progression or death
Overall survival | up to 60 months
  From the date of enrollment to the date of death or last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University shanghai cancer center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided